



## Contrasting Dosivent with Plus Flow Vu Spacer in Bronchial Hiperreactivity Patients

NCT: N/A

Date: 01/march/2022





## INFORMED CONSENT

| Contrasting Dosivent With Plus Flow Vu Spacer in Bronchial Hyperreactivity Patients | |
|---|---|
| I,been able to ask any questions regarding the study and understand that my participation in this study is volunta without any explanation. | , have read the patient information, ad have spoken to the study staff. I ary and can retire from it anytime I want, |
| I hereby give my consent to participate in this study: | |
| Participants name: | Investigator name: |
| Date and signature of participant: | Date and signature of investigatori |





Contrasting Dosivent With Plus Flow Vu Spacer in Bronchial Hyperreactivity Patients

This trial seeks comparison of bronchodilator testing between the use of Dosivent with Plus Flow Vu spacer in bronchial hyperreactivity patients.

For this to be done, two spirometries with bronchodilator testing in two different days are scheduled. One of the using the space chamber Dosivent and the other day using Aerochamber Plus Flow Vu spacer for 4 inhaled doses of Salbutamol. This test is done in Hospital Gregorio Marañon. Also, a satisfaction survery will be completed after using each of the devices.

As a participant, you are not gaining any immediate benefit for participating in this trial. Also, participating in this trial won't put you at any added risks from the ones of a regular scheduled bronchodilator testing.